CLINICAL TRIAL: NCT02826213
Title: Comparison of Two Techniques of Renal Pre-transplant Infusion on the Evolution of Renal Function in the Recipient: Multicentre Randomized Trial
Brief Title: Comparison of Two Techniques of Renal Pre-transplant Infusion on the Evolution of Renal Function in the Recipient
Acronym: RENOMAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRI14-JCV-RENOMAP
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Transplantation; Kidney
Keywords: Renal infusion; Renal infusion device

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kidney : perfusion device lifeport: Each donor (n=140) will provide one kidney for pulsatile perfusion.
  Interventions: Device: LifePort® perfusion device
- Kidney : perfusion device waves: Each donor (n=140) will provide one kidney for continuous perfusion.
  Interventions: Device: Waves perfusion device

INTERVENTIONS:
Device: LifePort® perfusion device — Renal Perfusion with LifePort® perfusion device
  Other Names: A
  Groups: Kidney : perfusion device lifeport
Device: Waves perfusion device — Renal Perfusion with Waves perfusion device
  Other Names: B
  Groups: Kidney : perfusion device waves

SUMMARY:
Comparison of two techniques of renal pre-transplant infusion on the evolution of renal function in the recipient: multicentre randomized trial

DETAILED DESCRIPTION:
Both machines differ in their operation: the LifePort® machine manufactured by the "Organ Recovery System (ORS)," says renal perfusion by maintaining a continuous perfusion pressure that is adjustable, while the Waves machine company "Medical Waters" assures infusion maintaining a controlled pulsatile flow.

Both machines are now available but the investigators currently have no study of whether an infusion type is superior to the other in terms of results on renal function recipients.

Study the impact of both types of infusion on renal function recipients evaluated in the early days of transplantation, at three months and one year after the transplant.

ELIGIBILITY:
RENAL Donors:

Inclusion Criteria:

* Deceased donor in brain-dead
* Donor presenting the expanded criteria of kidney removal (ECD criteria: elderly over 60 or aged 50 to 59 years and has two of the three following criteria: hypertension, stroke deaths, serum creatinine> 1.5 mg / dL)
* Possibility of both kidneys perfused machines
* Sampling of both kidneys, for two distinct recipients

Exclusion Criteria:

* none

RENAL recipients:

The grafts are addressed to transplant centers in France according to the distribution rules of the National Center of Distribution of transplants . (Pôle National de Répartition des Greffons (PNRG).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RENAL Donors and recipients
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | 3 months
  Rate of patients with a Glomerular Filtration Rate (GFR) calculated by the MDRD ≥ 45 ml / min / 1,73m² (considered normal in a renal graft) at 3 months post-transplantation (MDRD: Modification of Diet in Renal the Disease)

SECONDARY OUTCOMES:
Creatinine <250 mg / dL | 1 week
  Time for obtaining a serum creatinine <250 mg / dL and need for dialysis in recovery during the first seven days post transplant.
RFG | 1 month
  Absence of a recovery renal function at 1 month.
MDRD | 1 year
  Modification of Diet in Renal the Disease at 1 year
GSR | 1 year
  graft survival rate at 1 year.
Renal Biopsie results | 3 months
  Results of analyzes of kidney biopsies punctures to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe VENHARD, MD-PhD, Study Director — University Hospital, Tours
Locations (7):
- France (7):
  - Coordination Hospitalière de PMO , Pôle USSAR-Anestéthésie -Réa CHU-ANGERS, Angers
  - Coordination Hospitalière de PMO-Anestésiste -réanimateur, CHU-Bordeaux -GROUPE HOSPITALIER PELLEGRIN DAR I, Bordeaux
  - CHD-Vendée-Les Oudairies, La Roche-sur-Yon
  - Coordination des prélèvements d'organes et de Tissus- CHU-Limoges -CHU- DUPUYTREN, Limoges
  - Chirurgien-Chirurgie de la transplantation et d'Urologie, Pavillon V, Hôpital Edouard HERRIOT, Lyon
  - Coordination des prélèvements d'organes et de Tissus,CHU-NANTES, Nantes
  - Coordination des prélèvements d'organes et de Tissus Pôle Anesthésie-Réanimations,University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No